CLINICAL TRIAL: NCT04520451
Title: An Open Label, Two-Arm Study to Evaluate the Effect of Rilzabrutinib (PRN1008/SAR444671) on Safety and Disease Activity in ParticipantsWith IgG4-Related Disease
Brief Title: Open Label Two-Arm Study to Evaluate Rilzabrutinib in IgG4-Related Disease Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Principia Biopharma, a Sanofi Company (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT17125; PRN1008-017 (Other: Principia Biopharma Identifier); U1111-1260-3972 (Registry Identifier: ICTRP); 2022-002959-18 (EudraCT Number)
Record Dates: First submitted 2020-08-11; First posted 2020-08-20 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Immunoglobulin G4 Related Disease
Keywords: +IgG4; glucocorticoid; IgG4-RD; BTK; Bruton's
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rilzabrutinib + glucocorticoids (Experimental): Rilzabrutinib tablets, 400 mg twice daily from Week 0 to Week 12 plus glucocorticoids (20 to 40 mg/day prednisone equivalent tapered to 0 mg/day within 2 weeks on study)
  Interventions: Drug: rilzabrutinib; Drug: Glucocorticoids
- Glucocorticoids (Active Comparator): Glucocorticoids (20 to 40 mg/day prednisone equivalent tapered to 0 mg/day within 12 weeks on study)
  Interventions: Drug: Glucocorticoids

INTERVENTIONS:
Drug: rilzabrutinib — oral tablet
  Other Names: PRN1008/SAR444671
  Arms: Rilzabrutinib + glucocorticoids
Drug: Glucocorticoids — oral tablet or capsule

SUMMARY:
This is a Phase 2a, multi-center, open-label, two-arm study of approximately 25 patients with active IgG4-related disease (IgG4-RD). The two arms include (1) Experimental: rilzabrutinib with glucocorticoids and (2) Active Comparator: glucocorticoids only.

DETAILED DESCRIPTION:
4 weeks of screening, 12 weeks of main treatment, 12 weeks of cross-over (for GC-only group), 40 weeks of extension treatment and 4-week follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

* Be male or female with age ≥18 years.
* Have a clinical diagnosis of IgG4-RD.
* Be willing to taper off an equivalent prednisone dose of between 20-40 mg/day in 2 weeks.

Key Exclusion Criteria:

* Currently or within 6 months of screening taking rituximab, other B-cell depleting agents, or alkylating agents unless B cell concentrations have been demonstrated by flow cytometry to return to normal values (defined as 5 cells per cubic mm).
* History of solid organ transplant
* Positive at Screening for HIV, hepatitis B, hepatitis C, or TB
* Female patients who are pregnant or nursing.
* NOTE: Other Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-08-22 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who are without disease flare following the first dose of rilzabrutinib until the end of treatment | Up to 64 weeks
  Disease flare is defined as an increase in IgG4-RD responder index (RI) >2 or initiation of rescue treatment.
Incidence of SAE, AE leading to discontinuation and possible glucocorticoid-related AE | Up to 68 weeks
Number of participants with Potentially clinically significant abnormalities (PCSAs) for clinical laboratory tests, vital signs and ECG | Up to 68 weeks

SECONDARY OUTCOMES:
Proportion of participants with reduction from baseline IgG4-RD RI activity score by ≥2 points over time | At Week 52
Proportion of patients with an IgG4-RD RI activity score = 0 at over time | Up to 64 weeks
Level and change from baseline of each subclass of the serological markers over time | Up to 64 weeks
  serum protein electrophoresis to determine IgG subclasses and complement factors C3 and C4
Proportion of participants achieving reduction in baseline serum IgG4 level of 10% over time | Up to 64 weeks
Change from baseline in IgG4-RD RI over time | From baseline up to 64 weeks
Change from baseline in IgG4-RD damage, as recorded on the damage portion of the IgG4-RD RI over time | From baseline up to 64 weeks

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - Investigational Site Number 84019, Stanford, California
  - Investigational Site Number 84016, Boston, Massachusetts
  - Investigational Site Number 84018, Detroit, Michigan
  - Investigational Site Number 84030, New York, New York
  - Investigational Site Number 84036, Portland, Oregon
- Investigational Site Number 12403, Vancouver, Canada
- Investigational Site Number 25013, Marseille, France
- Investigational Site Number 38016, Milan, Italy
- Investigational Site Number 72415, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Wallace ZS, Zhang Y, Perugino CA, Naden R, Choi HK, Stone JH; ACR/EULAR IgG4-RD Classification Criteria Committee. Clinical phenotypes of IgG4-related disease: an analysis of two international cross-sectional cohorts. Ann Rheum Dis. 2019 Mar;78(3):406-412. doi: 10.1136/annrheumdis-2018-214603. Epub 2019 Jan 5. PMID 30612117